CLINICAL TRIAL: NCT07376655
Title: Effect of the Thrive AI Health App on Lifestyle Behaviors and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Thrive AI Health (Unknown)
Responsible Party: Principal Investigator, Melinda Irwin, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000040743
Record Dates: First submitted 2025-12-10; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Type 2; Overweight or Obesity
Keywords: Health app; Diet; Exercise; Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Motor Activity | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrive AI Health app (Experimental): Access to the Thrive AI Health app
  Interventions: Behavioral: App
- Wait list control (No Intervention)

INTERVENTIONS:
Behavioral: App — Access to the app during the 12 week period following randomization
  Arms: Thrive AI Health app

SUMMARY:
The goals of this randomized trial is to learn:

1. If the Thrive AI Health app will help adults improve their everyday habits (diet, exercise, and sleep).
2. How often participants will use the Thrive AI Health app to which they will have free access

The Thrive AI Health app uses artificial intelligence (AI) to give personalized advice. It is designed to help people eat better, exercise more, manage stress, and sleep well.

Researchers will compare changes in diet, exercise and sleep in participants using the app to those participants not using the app.

Participants will complete study questionnaires and an in-person visit at the beginning and end of the study.

DETAILED DESCRIPTION:
After consenting to participate in the study, adults who are overweight, have obesity, prediabetes, or type II diabetes will complete online questionnaires and attend an in-person visit.

The questionnaires measure:

Diet; Physical activity; Sleep quality; Quality of life

During the visit, the following will be measured or performed:

Height; Weight; Blood pressure; Blood sample collection; 6-minute walk test

Participants will then be randomly assigned to one of two groups:

1. Thrive AI Health app intervention group. The Thrive AI Health app uses artificial intelligence (AI) to give personalized advice. It is designed to help people eat better, exercise more, manage stress, and sleep well.
2. Wait-list control group

Those in the intervention group will be give a Fitbit which will by synched with the app.

After 12 weeks, participants will complete the questionnaires and clinic visit assessments again.

Following the 12-week assessments, those in the wait-list group will gain access to the Thrive AI Health app for 12 weeks and will complete online questionnaires at the 24-week mark.

When participants in the wait-list group gain access to the app, they will also start wearing a Fitbit, which will be linked to the app.

ELIGIBILITY:
Inclusion Criteria:

* Be at high risk for chronic disease defined as:

Body mass index (BMI)>25

BMI<=25 who are prediabetic or have type 2 diabetes

* Aged 40 years or older

Exclusion Criteria:

* Unable to walk

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Baseline to 12 weeks
  Self-reported minutes per week of moderate-vigorous-intensity physical activity will be estimated using the Modifiable Physical Activity Questionnaire. A higher number of minutes of moderate-vigorous-intensity physical activity per week means a better outcome.

SECONDARY OUTCOMES:
Healthy Eating Index | Baseline to 12 weeks
  Healthy Eating Index will be will be estimated using the self-reported food frequency questionnaire developed by Fred Hutchinson Cancer Center. The range for the Healthy Eating Index is 0-100. The higher number mean the better outcome
Sleep quality | Baseline to 12 weeks
  Self-reported sleep quality estimated using the Pittsburgh Sleep Quality Index (PSQI). Sleep will be assessed at baseline and 12-weeks using the PSQI, which is a widely used measure of subjective sleep disturbance; its validity and reliability have been established in various populations. Score range 0-21 with a lower score indicating better sleep.

OTHER OUTCOMES:
Body mass index | Baseline to 12 weeks
  Body mass index (wt/height squared) will be calculated using measured height and weight.
Aerobic capacity | Baseline to 12 weeks
  The widely used 6 minute walk test developed by the American Thoracic Society in 2002, will be used to assess aerobic capacity.
Physical quality of life score | Baseline to 12 weeks
  36-item Short Form Survey (SF-36) will be used to generate the Physical Component Summary (PCS). Using norm based scores, above 50 indicate a better-than-average physical health-related quality of life.
Mental quality of life score | Baseline to 12 weeks
  36-item Short Form Survey (SF-36) will be used to generate the Mental Component Summary (MCS). Using norm based scores, above 50 indicate a better-than-average mental health-related quality of life.